CLINICAL TRIAL: NCT06120270
Title: CeraFlex PFO Closure System Post-Market Clinical Follow-up Study: A Multi-center, Prospective, Observational, Post-market Study
Brief Title: CeraFlex PFO Closure System PMCF Study
Status: Recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT/TS/276I-2023-01
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Patent Foramen Ovale
Keywords: Lifetech; Patent Foramen Ovale; PFO; CeraFlex; CeraFlex PFO; CeraFlex PFO Closure System
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CeraFlex PFO Closure System — The Lifetech CeraFlex™ PFO occluder device is a percutaneous, transcatheter closure device for the non-surgical closure of Patent Foramen Ovale (PFO).

SUMMARY:
The purpose of this study is to compile real-world data on patient outcomes and evaluate the procedural success and performance of the CeraFlex™ PFO Closure System.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational, single-arm, open-label, post-market Study. The study device is the Lifetech CeraFlex PFO closure system, which is composed of a) CeraFlex PFO Occluder, and b) SteerEase Introducer. The PFO Closure System is indicated for the non-surgical closure of Patent Foramen Ovale (PFO), and the study objective is to collect real-world data on patient outcomes and evaluate the procedural success and performance of the CeraFlex PFO Closure System.

The estimated enrollment period is approximately 18 months, and each subject will followed 24 months post-procedure. The assessment schedule at discharge, 1-3 months follow-up, 6 months follow-up, 12 months follow-up, and 24 months follow-up.

Electronic Date Capture (EDC) System will be used for this Study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with indication(s) for PFO Occluder Closure in the Instruction For Use (IFU):

   1. Confirmed PFO by medical examinations;
   2. Associated with recurrent migraine/headache or TIA or cryptogenic stroke.
2. Patient characteristics consistent with the corresponding IFU & Device Size Selection:

   1. Measure the distance from the defect to the aorta root;
   2. Measure the distance from the defect to the superior vena cava (SVC) rim; select a device with the radius of the right disc that will not exceed the lesser of these two distances.
3. Patients who are willing to comply with all study procedures and be available for the duration of the study.
4. Patients or legally authorized representative(s) who are willing and capable of providing informed consent.

Exclusion Criteria:

1. Age <18 years or Age >85 years.
2. Patient with a history of ongoing Atrial Fibrillation (AF).
3. Patient with malignancy or other illness where life expectancy is less than 1 year.
4. Patient not covered by a social security scheme.
5. Patients who are participating in an investigational drug or device study currently.
6. Women of childbearing potential who are, or plan to become pregnant during the time of the study (method of assessment upon physician's discretion).
7. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
8. Any contraindication mentioned in the corresponding IFU：

   1. Patients known to have intracardiac thrombi, especially left atrial or left atrial appendage thrombi, demonstrated by echocardiography. Patients known to have a bleeding disorder, untreated ulcer, or any other contraindications to aspirin therapy unless another anti-platelet agent can be administered for 6 months.
   2. Anatomy in which the CeraFlexTM PFO device of the required size would interfere with intra-cardiac structure or intra-vascular structure, such as a pulmonary vein, or aorta root.
   3. Patients whose heart or vein size is too small to allow TEE probing or catheterization.
   4. Patients who are in the condition, e.g. active infection, which would cause them to be poor candidates for cardiac catheterization.
   5. Patients known to have sepsis within one month prior to implantation, or any systemic infection that cannot be successfully treated prior to device placement.
   6. Patients whose heart does not have enough tissue to secure the device.
   7. Patients with hypercoagulation disease.
   8. Any patient for whom the radius of the device is greater than the distance from the patent foramen ovale to the aortic root or superior vena cava.

      * No contraindications specified in the SteerEase introducer IFU.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PFO and need non-surgical closure of PFO.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Procedural success rate | Procedure/at discharge or 7 days post-procedure, whichever comes first
  Procedure success is defined as a composite of :
  1. absence of peri-procedural stroke-related events (ischemic stroke, cryptogenic stroke, or TIA), device embolization, cardiac or vascular perforation, or death, at discharge or 7 days post-procedure, whichever comes first;
  2. successful implantation of the device at the procedure.

SECONDARY OUTCOMES:
Residual shunt | At procedure, 6 months and 12 months post-implantation
  Residual shunt was classified on the basis of the estimated number of microbubbles detected in the left atrium within three cardiac cycles after appearance in the right atrium, as observed on cTTE/cTEE while the patient was at rest or during Valsalva procedure. The presence of 0 microbubbles was classified as no shunt, 1 to 5 microbubbles as small, 6 to 25 microbubbles as moderate, and more than 25 microbubbles as large.
Rate of stroke related events | From attempted procedure up to 24 months post-implantation
  Ischemic stroke, cryptogenic stroke, or TIA
Rate of Device Deficiencies | From attempted procedure up to 24 months post-implantation
  Including device malfunctions, failures, and non-conformances
Incidence of Serious Adverse Event | From attempted procedure up to 24 months post-implantation
  SAE
Incidence of death | From attempted procedure up to 24 months post-implantation
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Sandri, Dr, Principal Investigator — German Heart Center Leipzig
Locations (15):
- Germany (10):
  - Kardiologisch-Angiologische Praxis - Herzzentrum Bremen, Bremen
  - Heart Center Dresden, Dresden
  - Hospital Fürth, Fürth
  - Kath. Marienkrankenhaus gGmbH, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - German Heart Center Leipzig, Leipzig
  - Klinikum St. Georg gGmbH Leipzig, Leipzig
  - German Heart Center Munich, Munich
  - Herzzentrum Trier, Trier
  - University clinic Tübingen, Tübingen
- South Korea (5):
  - Yeungnam University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - ASAN Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Catholic University of Korea St. Vincent's Hospital, Suwon